CLINICAL TRIAL: NCT03072082
Title: Study of Curative Effect Evaluation of DanLou Tablet on Coronary Artery Disease Not Amenable to Revascularization on the Basis of Western Medicine Therapy
Brief Title: Curative Effect Evaluation of Danlou Tablet on Coronary Artery Disease Not Amenable to Revascularization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Li (Other)
Collaborators: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Jun Li, Director of Cardiology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLT-2016
Record Dates: First submitted 2017-02-22; First posted 2017-03-07 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease(CAD)
Keywords: coronary artery disease; revascularization; Danlou Tablet
MeSH Terms: conditions — Coronary Artery Disease | interventions — danlou tablet; Clopidogrel; Tablets; Atorvastatin; isosorbide-5-mononitrate; Metoprolol; Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danlou Tablet (Experimental): Danlou 0.3g tablet by mouth, 5 tablets three times daily for 6 months & conventional western medicine (including Aspirin Enteric-coated Tablets, Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet, Atorvastatin Calcium, Isosorbide Mononitrate Tab 20 MG, Metoprolol Tartrate Tab 25 MG, Trimetazidine Dihydrochloride Tablets)
  Interventions: Drug: Danlou Tablet; Drug: Aspirin Enteric-coated Tablets; Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet; Drug: Atorvastatin calcium; Drug: Isosorbide Mononitrate Tab 20 MG; Drug: Metoprolol Tartrate Tab 25 MG; Drug: Trimetazidine Dihydrochloride Tablets
- Danlou Tablet placebo (Placebo Comparator): Placebo Danlou 0.3g tablet by mouth, 5 tablets three times daily for 6 months & conventional western medicine (including Aspirin Enteric-coated Tablets, Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet, Atorvastatin Calcium, Isosorbide Mononitrate Tab 20 MG, Metoprolol Tartrate Tab 25 MG, Trimetazidine Dihydrochloride Tablets)
  Interventions: Drug: DanLou Tablet placebo; Drug: Aspirin Enteric-coated Tablets; Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet; Drug: Atorvastatin calcium; Drug: Isosorbide Mononitrate Tab 20 MG; Drug: Metoprolol Tartrate Tab 25 MG; Drug: Trimetazidine Dihydrochloride Tablets

INTERVENTIONS:
Drug: Danlou Tablet — Conventional western medicine & Danlou Tablet
  Arms: Danlou Tablet
Drug: DanLou Tablet placebo — Conventional western medicine & placebo (for Danlou Tablet)
  Arms: Danlou Tablet placebo
Drug: Aspirin Enteric-coated Tablets — 100 mg tablet, one tablet daily.
Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet — One tablet daily. (for patients who can't use aspirin)
  Other Names: Plavix
Drug: Atorvastatin calcium — 10 mg tablet, two tablets each night.
  Other Names: Lipitor
Drug: Isosorbide Mononitrate Tab 20 MG — One tablet two times daily.
  Other Names: Xinkang
Drug: Metoprolol Tartrate Tab 25 MG — 12.5 mg or 25 mg two times daily.
  Other Names: Metoprolol
Drug: Trimetazidine Dihydrochloride Tablets — 20 mg tablet, one tablet three times daily.
  Other Names: Vasorel

SUMMARY:
The purpose of this study is to determine whether Danlou Tablet is effective in the treatment of coronary artery disease not amenable to revascularization on the basis of western medicine therapy.

DETAILED DESCRIPTION:
The western medicine treatment for CAD not amenable to revascularization is limited. Danlou Tablet, a kind of Chinese patent medicine has been used for treating coronary artery disease in clinical practice in China for many years.

Danlou Tablet is applicable to "phlegm-stasis syndrome" in Traditional Chinese Medicine. According to recent studies, Danlou Tablet can reduce blood lipid level and myocardial necrosis area ,promote infarct healing in rats.And it can improve clinical symptoms of patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged between 45 and 75 years, diagnosed with sever CAD through coronary arteriography which shows that the left main coronary artery and three-vessel have sever diffuse stenosis, calcification or vascular ectasia, be in accordance with Traditional Chinese Medicine syndrome of "Qi deficiency and blood stasis syndrome" or "phlegm and stasis mu-tual obstruction syndrome".

Exclusion Criteria:

* Patients with severe valvular disease, congenital cardiomyopathy decompensation
* Patients with CAD complicated with severe multiple organ disease such as severe heart failure, severe lung, liver or renal dysfunction, peptic ulcer in active stage, or intracranial hemorrhage
* Patients that use high-dose steroids due to connective tissue disease
* Patients with serious infections
* Patients with malignant tumor
* Patients with hematopoietic diseases
* Pregnant or lactating women.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | Six months after randomisation
  Death caused by cardiovascular disease

SECONDARY OUTCOMES:
Ejection fraction percentage (EF%) | At baseline (before randomisation), and six months after randomisation
  One of Echocardiographic parameters
E/A ratio | At baseline (before randomisation), and six months after randomisation
  One of Echocardiographic parameters
C-reactive protein (CRP) | At baseline (before randomisation), and six months after randomisation.
  CRP in μg/L
B-type natriuretic peptide (BNP) | At baseline (before randomisation), and six months after randomisation.
  BNP in pg/mL
Hospital readmission rates | At baseline (before randomisation), and six months after randomisation.
  Hospital readmission rates due to coronary artery disease during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhao D. [Why dentists need to learn the epidemiological status and prevention strategy of coronary heart disease in China]. Zhonghua Kou Qiang Yi Xue Za Zhi. 2016 Jul;51(7):385-6. doi: 10.3760/cma.j.issn.1002-0098.2016.07.001. Chinese. PMID 27480425
- [Result] Zhu H, Luo XP, Wang LJ. [Evaluation on clinical effect of long-term shexiang baoxin pill administration for treatment of coronary heart disease]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2010 May;30(5):474-7. Chinese. PMID 20681275
- [Result] Zhou Z, Shen W, Yu L, Xu C, Wu Q. A Chinese patent medicine, Shexiang Baoxin Pill, for Non-ST-elevation acute coronary syndromes: A systematic review. J Ethnopharmacol. 2016 Dec 24;194:1130-1139. doi: 10.1016/j.jep.2016.11.024. Epub 2016 Nov 12. PMID 27847338
- [Result] Williams B, Menon M, Satran D, Hayward D, Hodges JS, Burke MN, Johnson RK, Poulose AK, Traverse JH, Henry TD. Patients with coronary artery disease not amenable to traditional revascularization: prevalence and 3-year mortality. Catheter Cardiovasc Interv. 2010 May 1;75(6):886-91. doi: 10.1002/ccd.22431. PMID 20432394
- [Result] Gupta S, Pressman GS, Morris DL, Figueredo VM. Distribution of left ventricular ejection fraction in angina patients with severe coronary artery disease not amenable to revascularization. Coron Artery Dis. 2010 Aug;21(5):278-80. doi: 10.1097/MCA.0b013e32833bdf53. PMID 20531008
- [Result] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Result] Wang L, Mao S, Qi JY, Ren Y, Guo XF, Chen KJ, Zhang MZ. Effect of Danlou Tablet () on peri-procedural myocardial injury among patients undergoing percutaneous coronary intervention for non-ST elevation acute coronary syndrome: A study protocol of a multicenter, randomized, controlled trial. Chin J Integr Med. 2015 Sep;21(9):662-6. doi: 10.1007/s11655-015-2284-1. Epub 2015 Jul 4. PMID 26142341
- [Result] Wang SH, Wang J, Li J. [Efficacy assessment of treating patients with coronary heart disease angina of phlegm and stasis mutual obstruction syndrome by Danlou tablet]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2012 Aug;32(8):1051-5. Chinese. PMID 23173251
- [Result] Chen J, Cai HW, Miao J, Xu XM, Mao W. [Danlou Tablet Fought against Inflammatory Reaction in Atherosclerosis Rats with Intermingled Phlegm and Blood Stasis Syndrome and Its Mechanism Study]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2016 Jun;36(6):703-8. Chinese. PMID 27491230